CLINICAL TRIAL: NCT03649139
Title: Effect and Underlying Immunological Mechanisms of Sublingual Immunotherapy in Seasonal Allergic Rhinitis: a Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Effect and Underlying Immunological Mechanisms of Sublingual Immunotherapy in Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Zhejiang Wolwo Bio-Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Luo Zhang, President, Beijing TongRen Hospital, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TR-SLIT-IMMUNO
Record Dates: First submitted 2018-08-02; First posted 2018-08-28 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Intervention Model Description: experiment:placebo=2:1
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artemisia annua (sweet sagewort) allergen extract drops (Active Comparator): Drug: sublingual immunotherapy drops
  Interventions: Drug: sublingual immunotherapy drops
- Placebo drops (Placebo Comparator): Drug: sublingual placebo drops
  Interventions: Drug: Placebo drops

INTERVENTIONS:
Drug: sublingual immunotherapy drops — artemisia annua (sweet sagewort) allergen extract drops
  Arms: artemisia annua (sweet sagewort) allergen extract drops
Drug: Placebo drops — sublingual placebo drops
  Arms: Placebo drops

SUMMARY:
Allergic rhinitis (AR) is a common Ig-E mediated disease of nasal mucosa, induced by an immunoglobulin E (IgE)-mediated reaction in the allergen-sensitized subjects, affecting 10% to 40% of the world population. AR could be divided into two kinds, perennial AR and seasonal AR (SAR). Allergen specific immunotherapy (AIT) is the only etiological treatment available for AR. Traditionally, AIT is divided into 2 types, subcutaneous immunotherapy (SCIT) and sublingual immunotherapy (SLIT), both of which are effective and safe alternatives.

The trial is a randomized, double-blind, placebo-controlled trial. 72 eligible SAR patients, who were sensitized to sweet sagewort (artemisia annua), were enrolled into the trial, followed by either a 32-week SLIT schedule, where the maintenance dose would be reached within 5 weeks, or placebo SLIT schedule. Standardized depot preparations of sweet sagewort (artemisia annua) extract (Zhejiang Wolwo Bio-pharmaceutical Co., Ltd., China ) were administered by means of sublingual drops.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 18 to 60 years (inclusive).
* With history of SAR for at least two years, with/without conjunctivitis and asthma
* Two or more nasal symptoms scores were ≥ 2 points during July - October in the last year.
* Sensitised to artemisia annua (specific IgE level ≥ 3.5 kilounit per liter).
* Patients who have been informed of the nature and aims of the study and have given their written consent, willing to comply with the protocol.
* Patients who are able to understand the information given and the consent and complete the daily record card.

Exclusion Criteria:

* Patients whose Humulus- or Artemisiifolia-specific immunoglobulin E (IgE) levels (ImmunoCAP) same as or higher than Artemisia-specific immunoglobulin E (IgE) level.
* Patients with oral diseases/ allergies within the run-in period.
* Patients accepted any kind of operations within 4 weeks of the run-in period.
* Patients applied for systemic glucocorticoids within 4 weeks in the run-in period.
* Patients with perennial AR.
* Patients with any nasal condition that could confound the results of the study (chronic rhinitis, chronic rhinosinusitis with/without polyps).
* Whatever the co-sensitization leading to clinically relevant AR, conjunctivitis or asthma likely to significantly change the symptoms of the patient throughout the study.
* Patients with comorbidity of severe asthma.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
change from baseline symptom scores at Week 16 | at baseline, Week 16
  Primary outcome is the assessment data from all patients whom will record on diary cards their symptom scores based on visual analog scales, ranging from 0(asymptomatic) to 3(most severe).

SECONDARY OUTCOMES:
Quality of life | at the pollen season of 2016, baseline, Week 16, Week 32, 6 months after discontinuation of treatment
  Assessment data from all patients whom will record on diary cards their quality-of-life measures for rhinitis(rhinoconjunctivitis quality of life questionnaire,RQLQ), including 28 questions, ranging from 0 (do not affect quality of life) to 6 (severely affect quality of life).
Medication scores | at the pollen season of 2016, baseline, Week 16, Week 32, 6 months after discontinuation of treatment
  Assessment data from all patients whom will record on diary cards their medication usage.
Immunologic Changes-IgE | at baseline, Week 16, Week 32
  Changes in total serum IgE, specific IgE levels in peripheral blood.
Immunologic Changes-M2 population | at baseline, Week 16, Week 32
  Changes in M2 population in peripheral blood and nasal secretion (Flow cytometry).
Change of symptom scores | at the pollen season of 2016, Week 16 and 6 months after discontinuation of treatment
  Assessment data from all patients whom will record on diary cards their symptom scores based on visual analog scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China